CLINICAL TRIAL: NCT00003423
Title: Non-Hodgkin's Lymphoma T Cell Protocol
Brief Title: Combination Chemotherapy in Treating Children With Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: United Kingdom Children's Cancer Study Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066443; UKCCSG-NHL-9503; EU-98012
Record Dates: First submitted 1999-11-01; First posted 2004-05-20 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2001-04

CONDITIONS: Lymphoma
Keywords: stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; stage I childhood large cell lymphoma; stage II childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma
MeSH Terms: conditions — Lymphoma; Dendritic Cell Sarcoma, Interdigitating | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Etoposide; Mercaptopurine; Methotrexate; Prednisolone; Thioguanine; Vincristine

INTERVENTIONS:
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: etoposide
Drug: mercaptopurine
Drug: methotrexate
Drug: prednisolone
Drug: thioguanine
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective for non-Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of different regimens of combination chemotherapy in treating children who have newly diagnosed non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether event-free survival for children with T-cell non-Hodgkin's lymphoma (NHL) can be improved by the addition of a third intensification block at 35 weeks. II. Determine biology and treatment response of T-cell NHL and T-cell acute lymphocytic leukemia when both are treated with an identical leukemia type protocol and receive a third intensification block. III. Improve the outcome for the 25% of children who are not in remission at eight weeks by the addition of a block of sustained intensification before high dose methotrexate and continuing treatment.

OUTLINE: Patients receive induction therapy on days 1-28. Patients receive supportive oral prednisolone daily for three doses during weeks 1-4, vincristine IV weekly for 5 weeks starting on day 1, asparaginase intramuscularly or subcutaneously three times a week beginning on day 4, and methotrexate intrathecally on days 1 and 8. Patients who meet certain criteria are given first intensification therapy beginning on day 29. Patients receive three doses of oral prednisolone, vincristine IV on day 1, daunorubicin IV over 6 hours on days 1 and 2, etoposide IV over 4 hours on days 1-5, cytarabine IV every 12 hours by bolus injection on days 1-5, oral thioguanine daily on days 1-5, and methotrexate intrathecally as in induction therapy. Patients are followed at 8 weeks. Those patients who experience remission receive a third intensification block at 35 weeks. All patients receive three methotrexate infusions followed by continuation therapy beginning at week 14. As continuation therapy, patients receive oral mercaptopurine daily, oral methotrexate weekly, vincristine IV every 4 weeks, oral prednisolone for 5 days every 4 weeks, and intrathecal methotrexate every 12 weeks beginning at week 23 until 100 weeks from the start of treatment. Continuation therapy will be interrupted at about week 20 for the second intensification therapy. For second intensification therapy, patients receive oral prednisolone daily for 5 days, a single dose of vincristine on day 1, daunorubicin IV over 6 hours on days 1 and 2, etoposide IV over 4 hours on days 1-5, bolus injections of cytarabine every 12 hours on days 1-5, oral thioguanine daily on days 1-5, and intrathecal methotrexate as in induction therapy. Continuation therapy re-starts at week 23. Patients who receive the third intensification therapy will begin at week 35. For the third intensification therapy, patients receive three doses of oral dexamethasone, IV vincristine on day 1 of weeks 35-38, subcutaneous asparaginase for 9 days during weeks 35-38, intrathecal methotrexate on day 1 of weeks 35 and 39, IV cyclophosphamide on day 1 of weeks 39 and 41, subcutaneous or IV cytarabine daily on days 1-4 of weeks 39- 42, and oral thioguanine daily during weeks 39-42. Continuation therapy re-starts at week 42/43. Some patients may receive radiotherapy during chemotherapy. Patients are followed every month for 1 year, every 2 months for the next year, every 6 months for the next 3 years, then annually thereafter.

PROJECTED ACCRUAL: Approximately 100 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed stage I, II, III, or IV T-cell non-Hodgkin's lymphoma No T-cell large anaplastic, peripheral T-cell lymphomas, or T-cell lymphoblastic leukemia No greater than 25% blasts in the bone marrow

PATIENT CHARACTERISTICS: Age: Under 15 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: No prior therapy

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 1995-05

CONTACTS AND LOCATIONS:
Overall Officials: Judith M. Chessells, MD, Study Chair — Institute of Child Health
Locations (1):
- Hospital for Sick Children NHS Trust, London, England, United Kingdom